CLINICAL TRIAL: NCT03722745
Title: Examine the Preliminary Effect of an Evidence-Based Practice (EBP) Consultation Model on Staff Fidelity to EBP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant recruitment due to high rates of staff turn over at three of the four recruitment sites
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-00792; 5K23MH104697-03 (NIH)
Record Dates: First submitted 2018-10-19; First posted 2018-10-29 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group 1 (Experimental): Juvenile offenders will attend 4-session Trauma Affect Regulation: Guide for Education & Treatment (TARGET) groups led by one or two juvenile staff members
  Interventions: Behavioral: TARGET
- study group 2 (Active Comparator): Juvenile offenders will receive treatment-as-usual (TAU).
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: TARGET — TARGET is manualized cognitive-behavioral treatment designed to help adolescents and adults with symptoms of posttraumatic stress
  Arms: Study group 1
Behavioral: TAU — It involves referral to an offsite community mental health provider with no attempt to control the treatment modality-type-quality (i.e., evidence-based-treatment or not).
  Arms: study group 2

SUMMARY:
Youth involved in the juvenile justice system report high rates of exposure to traumatic events (>90%) and posttraumatic stress disorder (PTSD; 20-50%). Although youth offenders are routinely assessed and referred for mental health services, few receive evidence-based interventions for PTSD. The current study evaluates an innovative approach to overcoming this problem: train front-line juvenile justice staff to deliver PTSD treatment groups. To determine the preliminary effectiveness and safety of PTSD groups delivered by juvenile justice staff, investigators will compare outcomes for youth offenders randomly assigned to receive evidence-based PTSD group treatment or treatment as usual (i.e., referral to community mental health clinic). Investigators hypothesize that PTSD groups led by justice staff will lead to significantly better youth outcomes (mental health symptoms, re-arrest) compared to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

Juvenile offender participants must

* be able to assent
* be between the ages of 13 and 17,
* currently involved with the local juvenile justice system (i.e., have an active court case),
* currently receiving services from one of the four participating agencies, and - meet DSM5 criteria for a full or partial diagnosis of Posttraumatic Stress Disorder (assessed during baseline eligibility screening with the eMINI-KID) or report moderate or greater PTSD symptoms on the UCLA PTSD-Reaction Index (score > 25).

Exclusion Criteria:

* unable to provide consent/assent
* Currently meet DSM5 criteria for Alcohol Use Disorder-Severe or any substance use disorders other than Cannabis or Nicotine (assessed with the eMINI-KID). This criterion is intended to exclude youth whose substance use is severe enough to require a higher level of care such as inpatient treatment;
* Currently meet DSM5 criteria for a psychotic disorder, pervasive developmental disorder, or other serious cognitive impairment (assessed with the eMINI-KID) that would prevent them from fully participating in the TARGET treatment groups;
* Report recent suicidal or homicidal ideation (i.e., past 6 months) or a past year suicide attempt unless the youth is currently receiving treatment from a licensed mental health professional (i.e., we will accept youth with recent SI/HI or past year suicide attempts if they are currently in treatment).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Youth PTSD symptoms | 8 Weeks
  University of California at Los Angeles (UCLA) Posttraumatic Stress Disorder Reaction Index-Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 version will be administered to assess youth symptom severity (range 0-124).
Youth PTSD re-arrest | 8 Weeks
  Number of times subject is arrested during study participation

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Branson, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared for any purpose.
  Researchers who provide a methodologically sound proposal will have access to the data.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date
Access Criteria: We will make the raw, de-identified final dataset publicly-available through the Inter-University Consortium for Political and Social Research (ICPSR) at the University of Michigan (http://www.icpsr.umich.edu). Investigators who wish to download our dataset will be required to first complete a standard data sharing agreement that includes: (1) a commitment to use the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. We are taking these steps to protect the confidentiality of study participants, given the restricted sample (justice-involved teens in NYC) and highly sensitive nature of the data (i.e., criminal record).